CLINICAL TRIAL: NCT02235480
Title: A Phase II Trial to Evaluate the Anti-psoriatic Efficacy and Tolerability of Tazarotene in a Gel Formulation in Patients With Mild to Moderate Nail Psoriasis - Parallel Group Comparison
Brief Title: Efficacy and Safety of Tazarotene Gel in Nail Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H 573 000 1307; 2013-004519-28 (EudraCT Number)
Record Dates: First submitted 2014-03-31; First posted 2014-09-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Nail Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tazarotene Gel (Experimental): once daily
  Interventions: Drug: Experimental Tazarotene Gel
- Placebo Gel (Placebo Comparator): once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Experimental Tazarotene Gel
  Arms: Tazarotene Gel
Drug: Placebo
  Arms: Placebo Gel

SUMMARY:
The aim of this study is to determine the efficacy and safety of topical application of the gel compared to placebo in nail psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Key inclusion criteria:
* Mild to moderate nail psoriasis on at least one fingernail

Exclusion Criteria:

Key exclusion criteria:

* any other skin condition, with a potential to affect the nails or to interfere with evaluation of the disease;
* history of hypersensitivity to retinoids or to other components of the trial medication
* topical treatment of nails with antipsoriatics in the 4 weeks preceding the treatment phase;
* systemic treatment of psoriasis within the three months before the treatment phase of the trial or during the trial
* intralesional steroid injection before the treatment phase of the trial
* phototherapy before the treatment phase of the trial;
* any chronic infection or condition capable of interfering with the conduct of the trial;
* evidence of drug or alcohol abuse;
* symptoms of a clinically significant illness that may influence the outcome of the trial in the four weeks preceding the treatment phase of the trial;
* participation in another clinical trial within the last 4 weeks prior to first treatment in this clinical trial;
* pregnancy or nursing;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
% reduction in the Nail Psoriasis Severity Index ( NAPSI ) | Day85

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 85

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Investigational site 3, Berlin
  - Investigational site 4, Berlin
  - Investigational 2, Hamburg
  - Investigational site 1, Hamburg